CLINICAL TRIAL: NCT01656564
Title: Clinical Outcomes in Persons With HIV Acquired Early in Life
Brief Title: Clinical Outcomes of People Who Acquired HIV in Early Life
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120157; 12-I-0157
Record Dates: First submitted 2012-07-31; First posted 2012-08-03 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: HIV
Keywords: HIV; Childhood; Antiviral Therapy; Cardiac; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Controls: Individuals with no known history of HIV
- Healthy Controls - Questionnaire Group: Individuals with no known history of HIV
- HIV: Individuals who acquired HIV in early life

SUMMARY:
Background:

- Long-term survival with the human immunodeficiency virus (HIV) is not well understood. Adults who were infected with HIV as children have lived with the virus for many years. However, the effect of HIV on this group of people has not been studied in depth. Researchers are interested in studying how HIV infection and the medicines used to treat it affect people who were infected early in life. They want to find out if there are any problems with how HIV-infected children grow and develop as adults, especially if they have developed heart problems. As part of this study, people with HIV will be compared with healthy volunteers.

Objectives:

- To study the effect of HIV infection and treatment on people who acquired HIV infection in early life.

Eligibility:

* Individuals at least 18 years of age who acquired HIV infection in early life.
* Healthy volunteers at least 18 years of age without HIV will serve as controls

Design:

* Participants will be screened with a physical exam and medical history. They will have regular study visits about once a year for up to 10 years to collect health information.
* Blood and urine samples will be collected to look at kidney and liver function.
* X-ray scans will be used to look at bone density and the amount of fat and muscle in the body.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Background:

* Antiretroviral therapy (ART) has altered the natural history of HIV disease in children.
* Long-term survivors of pediatric HIV infection offer a tremendous opportunity to understand the effects of HIV and ART health outcomes.
* A thorough understanding of the impact of HIV and ART on these long-term processes is extremely relevant as ART programs for HIV-infected children expand globally.

Objective:

- To explore the clinical outcomes and the impact of HIV infection and ART on a cohort with HIV infection acquired in early life

Eligibility:

* Individuals at least 18 years of age who acquired HIV infection in early life
* Healthy volunteers without HIV (greater than or equal to 18 years of age) will serve as controls

Design:

- Annual evaluations of health status, immune function and other health parameters related to HIV infection will be conducted.

ELIGIBILITY:
* INCLUSION CRITERIA:
* HIV positive participants

  * Known HIV infection, confirmed by laboratory testing and documented or believed to have been acquired during the first decade of life
  * Age greater than or equal to 18 years
* HIV negative controls

  * HIV negative, documented by a negative ELISA
  * Age greater than or equal to 18 years
  * Free of any major underlying medical disorder
  * Not currently pregnant

For Reproductive Health Sub-Study:

* HIV positive participants

  * Known HIV infection, confirmed by laboratory testing and documented or believed to have been acquired during the first decade of life
  * Age greater than or equal to 18 years
  * Capable of providing independent informed consent
* HIV negative controls

  * HIV negative, verified by a negative ELISA
  * Age greater than or equal to 18 years

For Healthy Volunteer, Questionnaire Group only

* Age >=18 years
* No known history of HIV

EXCLUSION CRITERIA:

Clinically significant condition or systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) which in the judgment of the Principal Investigator would compromise the patient s ability to tolerate this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected young adults; Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2012-08-27 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Health Status | End of Study
  vital status and health outcomes will be determined annually throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Hadigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.This is not an interventional study. This is a natural history study. Results are provided in aggregate in the form of published journal articles.

REFERENCES:
- [Background] Aepfelbacher JA, Chaudhury CS, Mee T, Purdy JB, Hawkins K, Curl KA, Dee N, Hadigan C. Reproductive and sexual health knowledge, experiences, and milestones in young adults with life-long HIV. AIDS Care. 2020 Mar;32(3):354-361. doi: 10.1080/09540121.2019.1679711. Epub 2019 Oct 22. PMID 31640401
- [Derived] Abd-Elmoniem KZ, Ishaq H, Purdy J, Matta J, Hamimi A, Hannoush H, Hadigan C, Gharib AM. Association of Coronary Wall Thickening and Diminished Diastolic Function in Asymptomatic, Low Cardiovascular Disease-Risk Persons Living with HIV. Radiol Cardiothorac Imaging. 2024 Apr;6(2):e230102. doi: 10.1148/ryct.230102. PMID 38573125
- [Derived] Sahagun SJ, Yeramosu T, Purdy JB, Reynolds JC, Hadigan CM. Associations Between Central Obesity and Lifelong Antiviral Therapy in Adults Living With HIV Acquired From Early Childhood. J Acquir Immune Defic Syndr. 2022 Feb 1;89(2):208-214. doi: 10.1097/QAI.0000000000002841. PMID 34693931
- [Derived] Aepfelbacher JA, Balmaceda J, Purdy J, Mattingly A, Zambell K, Hawkins K, Chairez C, Curl KA, Dee N, Hadigan C. Increased Prevalence of Hepatic Steatosis in Young Adults With Lifelong HIV. J Infect Dis. 2019 Jun 19;220(2):266-269. doi: 10.1093/infdis/jiz096. PMID 30852587
- [Derived] Unsal AB, Mattingly AS, Jones SE, Purdy JB, Reynolds JC, Kopp JB, Hazra R, Hadigan CM. Effect of Antiretroviral Therapy on Bone and Renal Health in Young Adults Infected With HIV in Early Life. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2896-2904. doi: 10.1210/jc.2017-00197. PMID 28531309
- [Derived] Mattingly AS, Unsal AB, Purdy JB, Gharib AM, Rupert A, Kovacs JA, McAreavey D, Hazra R, Abd-Elmoniem KZ, Hadigan C. T-cell Activation and E-selectin Are Associated With Coronary Plaque in HIV-infected Young Adults. Pediatr Infect Dis J. 2017 Jan;36(1):63-65. doi: 10.1097/INF.0000000000001354. PMID 27749650
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-I-0157.html